CLINICAL TRIAL: NCT07212218
Title: THE EFFECT OF HEALTH PROMOTION MODEL-BASED EDUCATION AND MOTIVATIONAL INTERVIEWS GIVEN TO PARENTS OF CHILDREN DIAGNOSED WITH TYPE 1 DIABETES ON DIABETES SELF-MANAGEMENT AND QUALITY OF LIFE
Brief Title: Health Promotion Model-Based Education and Motivational Interviewing for Parents of Children With Type 1 Diabetes
Acronym: HPM-T1D-MI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gözde EKŞİ, PhD Student, Public Health Nursing, Sağlık Bilimleri Üniversitesi, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBU-HSBE-T1D-01; 2023/3-3/10 (Other: Sağlık Bilimleri Üniversitesi Hamidiye Clinical Research Ethics Committe)
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus; Diabetes Self-Management; Quality of Life; Health Promotion Model (HPM); Motivational Interviewing (MI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Children with type 1 diabetes and their parents who voluntarily agree to receive the education will be included in the intervention group, while those who do not wish to participate in the training but agree to complete the assessments will be included in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Children with type 1 diabetes and their parents who voluntarily agree to participate will receive Health Promotion Model-based education sessions (~50-60 minutes) and motivational interviewing
  Interventions: Behavioral: Health Promotion Model-Based Education and Motivational Interviewing
- CONTROL Group (No Intervention): Children with type 1 diabetes and their parents in the control group will not receive any structured education or motivational interviewing during the study period. They will complete the same assessments (Diabetes Self-Management Scale, PedsQL Diabetes Module, and HbA1c data from medical records) at baseline and at 12 weeks. After study completion, they will be provided with the educational content

INTERVENTIONS:
Behavioral: Health Promotion Model-Based Education and Motivational Interviewing — Structured education sessions based on the Health Promotion Model will be delivered, followed by motivational interviewing techniques to enhance parental engagement and support diabetes management and quality of life.
  Arms: Intervention Group

SUMMARY:
This quasi-experimental study will aim to evaluate the effects of Health Promotion Model-based education and motivational interviewing on diabetes self-management and quality of life among parents of children diagnosed with type 1 diabetes. Eligible and voluntary parents will receive structured education sessions and motivational interviews designed to support diabetes management and improve quality of life. Outcomes will be assessed using validated questionnaires on diabetes self-management and quality of life, as well as HbA1c values obtained from patients' routine medical records. The study will examine whether parent-focused interventions can enhance diabetes management in children and families.

DETAILED DESCRIPTION:
This quasi-experimental study will be conducted to evaluate the effectiveness of Health Promotion Model-based education combined with motivational interviewing for parents of children diagnosed with type 1 diabetes. The theoretical framework will be based on Pender's Health Promotion Model, which emphasizes self-efficacy, perceived benefits, perceived barriers, and interpersonal influences in promoting health behaviors. Motivational interviewing techniques will be integrated to strengthen parental engagement and support behavioral change.

Participants will not be randomized into groups. Instead, parents who voluntarily accept to receive the education will form the intervention group, while those who prefer not to participate in the training but agree to complete the evaluation will form the control group. The intervention will consist of structured education sessions lasting approximately 50-60 minutes, delivered in the pediatric endocrinology clinic setting, followed by motivational interviews.

Data will be collected at baseline and 12 weeks after the intervention. The evaluation will include validated measurement tools such as the Diabetes Self-Management Scale, the Pediatric Quality of Life Inventory (PedsQL) Diabetes Module, and HbA1c values obtained from patients' routine medical records. The study is anticipated to provide evidence on the effectiveness of Health Promotion Model-based education and motivational interviewing in strengthening parental support, thereby improving diabetes self-management in children with type 1 diabetes and enhancing quality of life for both children and their families.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 8-12 years with type 1 diabetes diagnosed for ≥ 1 year HbA1c ≥ 7% Using insulin pen for treatment Able to read and write Living in Istanbul No intellectual disability No other chronic disease Parent able to communicate by phone and use social media apps (e.g., WhatsApp, Zoom) Both child and parent willing to participate

Exclusion Criteria:

* sychiatric disorder diagnosis Type 1 diabetes diagnosis < 1 year Using insulin pump or other treatment methods Having another type of diabetes Not in the 8-12 age range Illiteracy (child or parent) Presence of another chronic disease Parent unable to use phone or social media apps Child and/or parent unwilling to participate

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management Scale | Baseline and 12 weeks after intervention
  The Diabetes Self-Management Scale will be used to assess self-management skills of children with type 1 diabetes. Scores will be compared between baseline and post-intervention assessments.
Change in Quality of Life (PedsQL Diabetes Module) | Baseline and 12 weeks after intervention
  Quality of life in children with type 1 diabetes will be assessed using the PedsQL Diabetes Module. Scores will be compared between baseline and post-intervention.

SECONDARY OUTCOMES:
Change in HbA1c (%) | Baseline and 12 weeks after intervention
  HbA1c values will be obtained from patients' routine clinical records measured by endocrinologists

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Ekşi, PhD Candidate, Principal Investigator — University of Health Sciences, Hamidiye Institute of Health Sciences
Locations (1):
- Umraniye Training and Research Hospital, Pediatric Endocrinology Clinic, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns. Only aggregate data will be reported.

REFERENCES:
- See also: This article reports the development and validation of the PedsQL Diabetes Module, which will be used in this study to assess quality of life in children with type 1 diabetes. — https://pubmed.ncbi.nlm.nih.gov/12610013/
- See also: The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control — https://pubmed.ncbi.nlm.nih.gov/23937988/
- See also: This article provides the 2024 American Diabetes Association Standards of Care in Diabetes, which serve as evidence-based clinical guidelines for diabetes management and are referenced in the study protocol. — https://pubmed.ncbi.nlm.nih.gov/38119244/